CLINICAL TRIAL: NCT00717535
Title: Investigation of the Total Nucleated Cell Yield of Cord Blood Units Collected From African-American Donors in Correlation With Gestational and Other Health Variables
Brief Title: Studying Umbilical Cord Blood From African-American Donors
Status: Withdrawn | Type: Observational
Why Stopped: Funding unavailable
Sponsor: Barbara Ann Karmanos Cancer Institute (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CDR0000598111; P30CA022453 (NIH); WSU-C-2933; WSU-W81XWH-05-1-0266; WSU-024405MP4E (Other: Wayne State University - Human Investigation Committee); WSU-0505001823 (Other: Wayne State University - Human Investigation Committee)
Record Dates: First submitted 2008-07-16; First posted 2008-07-17 (Estimated); Last update posted 2013-04-29 (Estimated); Status verified 2013-04

CONDITIONS: Health Status Unknown
Keywords: health status unknown
MeSH Terms: interventions — Cryopreservation

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: None Retained — Cord blood unit (CBU)will be collected in utero and transported to the Stem Cell Processing Laboratory. The volume of the CBU will be measured and cell count will be obtained.
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: cryopreservation
Other: questionnaire administration
Other: study of socioeconomic and demographic variables

SUMMARY:
RATIONALE: Studying umbilical cord blood in the laboratory and gathering information about current and previous pregnancies from African-American umbilical cord blood donors may help doctors learn more about the umbilical cord blood of these donors.

PURPOSE: This clinical trial is looking at umbilical cord blood from African-American donors.

DETAILED DESCRIPTION:
OBJECTIVES:

* To correlate the total nucleated cell yield of cord blood units from African-American cord blood donors with gestational history, maternal history, and delivery information.

OUTLINE: This is a multicenter study.

Donors complete questionnaires about their demographics, maternal history, gestational history, and delivery. Cord blood units (CBU) are collected in utero and transported to the Stem Cell Processing Laboratory where they are evaluated for CBU volume and cell count (i.e., total nucleated cell yield) and cryopreserved. The study results will then be used to devise future interventional strategies to improve the yield of nucleated cells of CBU.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* African-American participant in the National Marrow Donor Program cord blood collection protocol C-2844
* Recruited from the Labor and Delivery Suites of the Detroit Medical Center or its affiliated sites

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* Not specified

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: African American cord blood donors
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2005-08; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Correlation between total nucleated cell yield of cord blood units and gestational history, maternal history, and delivery information | Within a year
Improvement in total nucleated cell yield of cord blood units from African-American donors | Within a year

CONTACTS AND LOCATIONS:
Overall Officials: Voravit Ratanatharathorn, MD, Principal Investigator — Barbara Ann Karmanos Cancer Institute